CLINICAL TRIAL: NCT04666116
Title: Changes in Viral Load in Patients With COVID-19 Disease After Dietary Supplementation With Probiotics: A Randomized Clinical Trial
Brief Title: Changes in Viral Load in COVID-19 After Probiotics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Sagunto (Other)
Collaborators: Biopolis S.L. (Industry); Laboratorios Heel España (Unknown)
Responsible Party: Principal Investigator, Xavier Cortés, Digestive specialist from the Internal Medicine Service, Hospital de Sagunto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HdeSagunto
Record Dates: First submitted 2020-04-25; First posted 2020-12-14 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: COVID-19
Keywords: COVID-19; probiotic supplementation; GASTEEL PLUS
MeSH Terms: conditions — COVID-19 | interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Randomized, single blind clinical trial
Who Masked: Outcomes Assessor
Masking Description: Computerized randomization based on a single sequence based on the latest issue in the patient's medical history
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID-19 patients no dietary administration (No Intervention): Only medication agreed by the hospital committee
- COVID-19 patients with dietary administration (Experimental): Medication agreed by the hospital committee and nutritional supplement.
  Interventions: Dietary Supplement: Dietary supplementation in patients with covid disease admitted to hospital

INTERVENTIONS:
Dietary Supplement: Dietary supplementation in patients with covid disease admitted to hospital — Dietary supplementation in patients with covid disease admitted to hospital
  Arms: COVID-19 patients with dietary administration

SUMMARY:
The main objective of the study is to evaluate the capacity of a novel nutritional supplement intervention including strains from the species Bifidobacterium longum, Bifidobacterium animalis subsp. Lactis and Lactobacillus rhamnosus, plus vitamin D, zinc and seleniumt) (immune system enhancer, antioxidant and anti-inflammatory capacity) to decrease the viral load by nasopharyngeal smear in patients admitted for COVID-19 coronavirus disease.

DETAILED DESCRIPTION:
1. Study hypothesis: Through the administration of specific probiotics, the immune response against the coronavirus COVID-19 could be stimulated, being able to decrease its viral load and secondary symptomatology.

   There is a different way to attack a harmful microorganism. It is based on the existence in its habitat of a whole complex network of other microorganisms, our microbiota, which prevents the development, growth and feeding of that microorganism, either by competition of space, food, or immune effects. In COVID-19 patients, intestinal dysbiosis has been described, specifically observing the decrease of species considered as probiotics of the genera Lactobacillus and Bifidobacterium. The current study proposes the testing of the novel nutritional supplement to potential the patient's immune system and balances the damaged microbiota. This product contains species from the genera described as affected in the COVID-19 infection. Moreover, the strains selected showed an anti-inflammatory and antioxidant effect, and capacity for stimulation of the immune system in previous assays. All three strains have the GRAS status recognized by the FDA and are on the EFSA QPS list. The product also contains vitamin D, zinc and selenium, three powerful inducers of the immune response. It is a safe product according to WHO criteria. In addition, it can be effective despite the administration of antibiotics, due to postbiotic activity, reducing the risk of sepsis described in this type of patient. In order to monitor the effects of treatment with the functional product, a follow-up will be made by means of consultation regarding the evolution of the patient's condition. On the other hand, we will try to correlate this state with the viral load present in serum and pharyngeal-nasal scraping.
2. PRIMARY AND SECONDARY OBJECTIVES

Main objective: The main objective of the study is to evaluate the capacity of the novel nutritional supplement (immune system enhancer, antioxidant and anti-inflammatory capacity) to decrease the viral load by nasopharyngeal smear in patients admitted for COVID-19 coronavirus disease. The Patient will follow the medication agreed by the Hospital committee during all the process.

Secondary objectives: Monitoring of changes, in patients admitted by COVID-19+, of the following parameters at admission and prior to discharge:

* Hospital stay (days). Stay in Intensive Care Unit (days)
* Clinical indicators: Respiratory rate, body temperature, number of bowel movements and consistency. Abdominal pain. Nausea and vomiting. Sat02.
* Type of respiratory support on day 5 of admission: ambient air (none), nasal mask, ventimask, reservoir, non-invasive mechanical ventilation (NIV), orotracheal intubation.
* Analytical parameters at admission and discharge: Total lymphocytes, Hemoglobin, Ferritin, Neutrophils, Urea/Creatinine, C-reactive protein, LDH, D-dimer, AST/ALT, Platelets.
* Determination of the incidence of mortality in the patient cohort and comparison with that described in the literature.

  3. PRIMARY AND SECONDARY STUDY VARIABLES

  3. 1. Primary study variable
* Viral load during the period of admission to the nasopharyngeal smear.

  3. 2. Secondary study variables
* Hospital stay (days). Stay in Intensive Care Unit (days).
* Clinical indicators on admission and every 48 hours thereafter: Respiratory rate, oxygen saturation, body temperature, number of bowel movements and consistency. Abdominal pain. Nausea and vomiting.
* Type of respiratory support on the 5th day of admission: ambient air (none), nasal glasses, ventimask, reservoir, non-invasive mechanical ventilation (NIV), orotracheal intubation.
* Mortality.
* Analytical parameters at day 0 and at hospital discharge: Total lymphocytes, ferritin, hemoglobin, neutrophils, urea/creatinine, C-reactive protein, IL-6, LDH, D-dimer, AST/ALT, platelets
* Appearance of side effects.

  4. MATERIAL AND METHODS

4.1. Study design Randomized clinical trial with a clinical intervention of prescription of functional novel nutritional supplement. The expected duration is 3 months in all patients presenting symptoms of infection by COVID-19 or COVID+.

Serum viral load will be analyzed by rt-qPCR (reverse transcriptase quantitative Polymerase Chain Reaction) at the beginning of the patient's admission and every 48 hours until remission of the infection and pharyngeal-nasal exudate.

The patient medicated according to hospital protocol will also be given a daily dose (one sachet) until remission of the illness or for one month.

4.2. Sample size of the study According to GRANMO Sample Size Calculator (Version 7.12 April 2012) Accepting an alpha risk of 0.15 and a beta risk of 0.3 in a bilateral contrast, 48 subjects in the first group and 48 in the second are required to detect the difference between two proportions as statistically significant, than for group 1 (intervention group) it is expected to be 0.5 and group 2 0.7. A follow-up loss rate of 5% has been estimated. The ARCOSENE approach has been used.

4.3. Statistical plan Quantitative variables will be expressed as mean and standard deviation assuming normal distribution based on the central limit theorem.

Qualitative variables will be expressed as frequencies with their 95% confidence intervals. Qualitative variables will be compared using the Chi-square test.

Quantitative variables will be compared using the Student T test. In order to evaluate the impact of the intervention on the evolution of the disease by COVID-19, on average stay, clinical variables and qualitative and quantitative analyses, a multivariate analysis will be carried out, in which it will be controlled by different variables that could act as factors of confusion (age, sex, type of disease, severity of the disease on admission, other diseases that could affect the evolution, medical treatment, previous surgeries, etc.)

4.4. Planning the physical-sample drawing Main evaluation criteria: These patients will have their surgery performed pharyngeal-nasal smear on day 0 and day 5 of hospital admission.

Viral load testing and cytokines: In the samples, the viral load will be determined by rt-qPCR, in hospital services. Cytokines shall be measured at the indication of the physician when deemed appropriate.

5. ETHICAL ASPECTS TAKEN INTO ACCOUNT IN THE STUDY PROTOCOL

5.1 Ethical conduct of the study

The study will be carried out in accordance with the following guidelines:

* Local ethical standards.
* European directives on the protection of human subjects in research.
* Declaration of Helsinki.
* The study will be conducted in strict accordance with the international ethical recommendations for human research and clinical trials set out in the Declaration of Helsinki, and in accordance with the recommendations of the Ministry of Health on clinical trials.
* Recommendations of the European Network of Pharmacoepidemiology and Pharmacovigilance Centres
* GMP recommendations.
* Other relevant guidelines, laws or regulations applicable in each country and in the Valencian Community As it is a research project with a nutritional supplement, it is not considered a medicine or a health product, and therefore the Biomedical Research Law applies to it and not the EECC RD 1090/2015. Therefore, there is no need for authorization by the AEMPS (State Agency for Medicines) or by the Conselleria de Sanitat.

The study protocol will be submitted for prior approval to the Hospital de Sagunto IRB.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age admitted to the Internal Medicine Unit of Sagunto Hospital, for illness due to infection secondary to COVID-19 during the study period.
* To be willing and able to sign the informed consent to participate

Exclusion Criteria:

* Not meeting any of the inclusion criteria.
* Present allergy to any of the components of the nutritional supplement Gasteel Plus.
* Not being able to ingest anything by mouth, either by dysphagia or by prescription.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Viral load during the period of admission to the nasopharyngeal smear. | 1 year
  The main objective of the study is to evaluate the capacity of the nutritional supplement (immune system enhancer, antioxidant and anti-inflammatory capacity) to decrease the viral load by nasopharyngeal smear in patients admitted for COVID-19 coronavirus disease

SECONDARY OUTCOMES:
Clinical indicators on admission and every 48 hours thereafter | 1 year
  non-invasive mechanical ventilation (NIV) intervention, (yes or not)
Analytical parameters | 1 year
  IL-6 initial point. (pg/mL)
Mobility | 1 year
  Hospital stay (days) and Stay in Intensive Care Unit (days).
Microbiome analysis in feces | 1 year
  Generation of a collection of PCRs products individually labelled from the hypervariable region of the 16s rRNA. After QC, each sample will be PCR amplified using a specific combination of primers specially designed and adapted for massive sequencing to capture the hypervariable region V3-V4 of the bacterial 16s rRNA (Klindworth et al. 2013). Sequencing in a illumina Miseq equipment.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital de Sagunto, Sagunto, Valencia
  - Hospital de Sagunto, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Reino-Gelardo S, Palop-Cervera M, Aparisi-Valero N, Espinosa-San Miguel I, Lozano-Rodriguez N, Llop-Furquet G, Sanchis-Artero L, Cortes-Castell E, Rizo-Baeza M, Cortes-Rizo X. Effect of an Immune-Boosting, Antioxidant and Anti-Inflammatory Food Supplement in Hospitalized COVID-19 Patients: A Prospective Randomized Pilot Study. Nutrients. 2023 Apr 1;15(7):1736. doi: 10.3390/nu15071736. PMID 37049576